CLINICAL TRIAL: NCT00565292
Title: A Study of MK0859 in Patients With Primary Hypercholesterolemia or Mixed Hyperlipidemia (MK-0859-011)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-011; 2007_655
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Hypercholesterolemia; Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — anacetrapib

INTERVENTIONS:
Drug: MK0859

SUMMARY:
This is a study to assess the safety, efficacy, and tolerability of MK0859 in patients with primary hypercholesterolemia (large amounts of cholesterol in the blood) or mixed hyperlipidemia (high levels of LDL cholesterol, triglycerides, and low levels of HDL cholesterol in blood) This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years of age
* Patient can be on a stable diet for the study
* Patient has a stable weight for more then 6 weeks before the study and has not participated in a weight loss program

Exclusion Criteria:

* Patient has chronic heart failure or a history of heart disease
* Patient has blood, digestive, or central nervous system disorders
* Patient is pregnant or nursing
* Patient is HIV positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Krishna R, Anderson MS, Bergman AJ, Jin B, Fallon M, Cote J, Rosko K, Chavez-Eng C, Lutz R, Bloomfield DM, Gutierrez M, Doherty J, Bieberdorf F, Chodakewitz J, Gottesdiener KM, Wagner JA. Effect of the cholesteryl ester transfer protein inhibitor, anacetrapib, on lipoproteins in patients with dyslipidaemia and on 24-h ambulatory blood pressure in healthy individuals: two double-blind, randomised placebo-controlled phase I studies. Lancet. 2007 Dec 8;370(9603):1907-14. doi: 10.1016/S0140-6736(07)61813-3. PMID 18068514